CLINICAL TRIAL: NCT01589497
Title: Essentiality of Isoniazid in Tuberculosis Therapy
Brief Title: Essentiality of INH in TB Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5307; 1U01AI068636 (NIH)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin; Isoniazid; Pyrazinamide; Ethambutol; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RHZE-RHZE (Active Comparator): Participants were administered rifampin-isoniazid-pyrazinamide-ethambutol (RHZE) from Day 1 to Day 14.
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol
- RHZE-RZE (Active Comparator): Participants were administered RHZE from Day 1 to Day 2, then rifampin-pyrazinamide-ethambutol (RZE) from Day 3 to Day 14.
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol
- RHZE-RMZE (Active Comparator): Participants were administered RHZE Day 1 to Day 2 and rifampin-moxifloxacin-pyrazinamide-ethambutol (RMZE) from Day 3 to Day 14.
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Moxifloxacin
- RZE-RZE (Active Comparator): Participants were administered only RZE from Day 1 through Day 14.
  Interventions: Drug: Rifampicin; Drug: Pyrazinamide; Drug: Ethambutol

INTERVENTIONS:
Drug: Rifampicin — Participants with body weight </= 50kg were administered one 450 mg tablet orally once daily. Participants with body weight >50kg were administered one 600 mg tablet orally once daily.
Drug: Isoniazid — Participants were administered three 100 mg tablets or one 300 mg tablet once daily.
  Arms: RHZE-RHZE; RHZE-RMZE; RHZE-RZE
Drug: Pyrazinamide — Participants with a body weight of 40-55 kg were administered two 500 mg tablets orally once daily. Participants with a body weight of 56-75 kg were administered three 500 mg tablets orally once daily. Participants with a body weight of 76-90 kg were administered four 500 mg tablets orally once daily.
Drug: Ethambutol — Participants with a body weight of 40-55 kg were administered two 400 mg tablets orally once daily. Participants with a body weight of 56-75 kg were administered three 400 mg tablets orally once daily. Participants with a body weight of 76-90 kg were administered four 400 mg tablets orally once daily.
Drug: Moxifloxacin — Participants were administered one 400 mg tablet orally once a day.
  Other Names: Avelon
  Arms: RHZE-RMZE

SUMMARY:
Tuberculosis (TB) disease is caused by bacteria that have infected the lung. TB bacteria are very small living agents that are spread by coughing and can be killed by taking TB drugs. To kill these TB bacteria TB patients have to take a combination of four drugs for 2 months and then two drugs for a further 4 months. During the first 2 months patients take rifampicin, isoniazid, ethambutol, and pyrazinamide. After that patients take only isoniazid and rifampicin for a further 4 months, making a total of 6 months therapy.

In A5307 the investigators wanted to test a new combination of drugs to see if the investigators could treat TB faster in the future.

Studies in animals have suggested that one of the four drugs, isoniazid, only works for a few days and may not be needed after the first two doses of TB treatment to kill the TB bacteria. After that its effects wear off to the point that it may even interfere with the other drugs. The investigators wanted to see if stopping isoniazid early, or using moxifloxacin, a different drug, instead could treat TB faster. This study was the first time that this type of regimen without isoniazid had been tested in humans. If the investigators could show that isoniazid stops working after a few days, the investigators could then try to see if they could possibly make a better tuberculosis treatment in the future.

DETAILED DESCRIPTION:
This was a Phase IIa open label, randomized clinical trial comparing the early bactericidal activity (EBA) of four anti-tuberculosis regimens. Participants with acid fast bacilli (AFB) smear-positive pulmonary tuberculosis were hospitalized from screening through Day 15 of the study, during which time, sputum, blood, and urine were collected. Participants returned to the clinic on Day 28 for the final visit. The study duration was 29 days.

The purpose of the study was to estimate the primary outcome within each study arm and the study was not designed for between arm comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Absence of HIV-1 infection within 30 days prior to study entry OR
* HIV-1 infection
* Sputum positive for acid fast bacilli (AFB) by smear-microscopy ≥1+ on the WHO/IUALTD scale within 1 day prior to study entry.
* Isoniazid and rifampin sensitivity, based on Hain GenoType MTBDR Plus assay performed within 7 days prior to study entry.
* Body weight: 40 kg to 90 kg, inclusive
* Age ≥ 18 years at study entry.
* Certain laboratory values, as defined in the protocol, obtained within 30 days prior to entry
* For HIV-positive candidates only: CD4+ cell count of > 200 cells/mm^3, determined within 7 days prior to study entry at a DAIDS approved laboratory.
* For females of reproductive potential, negative serum or urine pregnancy test within 7 days prior to entry.
* Female participants who are participating in sexual activity that could lead to pregnancy must agree to use one reliable non-hormonal form of contraceptive (ie, condoms, with a spermicidal agent; a diaphragm, or cervical cap with spermicide; or an IUD) while receiving study medications.
* Radiographic findings consistent with pulmonary TB from a chest x-ray performed within 14 days prior to entry.
* Ability and willingness of study candidate or legal guardian/representative to provide informed consent.
* Willingness to be hospitalized for approximately 3 weeks.
* Ability to provide at least 10mL of sputum during an overnight collection prior to study entry.

NOTE: Candidates who do not produce an overnight sputum sample of sufficient quality and quantity will be considered screen failures. However, if a candidate's failure to produce sufficient sputum appears to be due to poor technique rather than low volume of sputum production, this evaluation may be repeated.

Exclusion Criteria:

* Receipt of INH prophylaxis or any tuberculosis therapy within 7 days prior to study entry or for more than 7 cumulative days in the last 6 months, or receipt of any fluoroquinolone in the 1 month prior to entry.
* Currently on anti-retroviral treatment (ART), has been on ART within 30 days, or is expected to initiate ART within 2 weeks after study entry.
* Breastfeeding.
* Known intolerance to any of the study drugs.
* Resistance to rifampicin determined by GeneXpert within 7 days prior to study entry.
* Known history of resistance to isoniazid or rifampin or known close exposure (i.e., household exposure) to someone with MDR TB or known study candidate default on previous TB treatment (ie, the study candidate was diagnosed with TB, started TB treatment but did not complete that treatment).
* Known allergy to any fluoroquinolone antibiotic.
* History of prolonged QT syndrome or a QTc of > 450 ms (using Fridericia's correction)..
* Current or planned therapy with quinidine, procainamide, amiodarone, sotalol, or ziprasidone during the 2 weeks of on-study tuberculosis treatment.
* Current or prior diagnosis of pulmonary silicosis.
* Advanced disease as defined by Karnofsky score ≤ 70 at screening.
* Any of the following current comorbidities, complications, or underlying medical conditions:

  * poorly controlled diabetes, as determined by the site investigator
  * currently uncontrolled hypertension (ie, requiring acute medical treatment or immediate hospitalization)
  * miliary TB
  * neurological TB (including TB of the spine, TB meningitis)
  * peripheral neuropathy ≥ Grade 2 according to the December 2004 (Clarification, August 2009) Division of AIDS (DAIDS) Toxicity Table, within 90 days prior to study entry
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Estimated overnight sputum production of < 10 mL.
* Requirement for concomitant medications that may potentially interact with study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-06-30; Primary Completion 2016-01-28 (Actual); Study Completion 2016-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bishai, MD, PhD, Study Chair — Johns Hopkins Center for TB Research; Andreas Diacon, MD, PhD, Study Chair — TASK Applied Science CRS
Locations (2):
- South Africa (2):
  - University of Cape Town Lung Institute (UCTLI) CRS (31792), Cape Town, Western Cape
  - TASK Applied Science CRS (31718), Bellville

REFERENCES:
- [Background] The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009).
- [Derived] Diacon A, Miyahara S, Dawson R, Sun X, Hogg E, Donahue K, Urbanowski M, De Jager V, Fletcher CV, Hafner R, Swindells S, Bishai W. Assessing whether isoniazid is essential during the first 14 days of tuberculosis therapy: a phase 2a, open-label, randomised controlled trial. Lancet Microbe. 2020 Jun;1(2):e84-e92. doi: 10.1016/s2666-5247(20)30011-2. Epub 2020 Jun 8. PMID 33834177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at two AIDS Clinical Trials Units in South Africa. Recruitment occurred between June 30, 2015 (date of first participant was randomized) and January 13, 2016 (date of last participant was randomized).
Pre-assignment Details: 69 were randomized 1:1:1:1 to 4 treatment arms. Among the 69 participants, 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Groups:
- RHZE-RHZE: Participants were administered RHZE from Day 1 to Day 14. Rifampicin: Participants with body weight </= 50kg were administered one 450 mg tablet orally once daily; with body weight >50kg were administered one 600 mg tablet orally once daily.
  Isoniazid: Participants were administered three 100 mg tablets or one 300 mg tablet once daily.
  Pyrazinamide: Participants with a body weight of 40-55 kg were administered two 500 mg tablets orally once daily; with a body weight of 56-75 kg were administered three 500 mg tablets orally once daily; with a body weight of 76-90 kg were administered four 500 mg tablets orally once daily.
  Ethambutol: Participants with a body weight of 40-55 kg were administered two 400 mg tablets orally once daily; with a body weight of 56-75 kg were administered three 400 mg tablets orally once daily; with a body weight of 76-90 kg were administered four 400 mg tablets orally once daily.
- RHZE-RZE: Participants were administered RHZE from Day 1 to Day 2, then RZE from Day 3 to Day 14.
  Rifampicin: Participants with body weight </= 50kg were administered one 450 mg tablet orally once daily; with body weight >50kg were administered one 600 mg tablet orally once daily.
  Isoniazid: Participants were administered three 100 mg tablets or one 300 mg tablet once daily.
  Pyrazinamide: Participants with a body weight of 40-55 kg were administered two 500 mg tablets orally once daily; with body weight of 56-75 kg were administered three 500 mg tablets orally once daily; with a body weight of 76-90 kg were administered four 500 mg tablets orally once daily.
  Ethambutol: Participants with a body weight of 40-55 kg were administered two 400 mg tablets orally once daily; with a body weight of 56-75 kg were administered three 400 mg tablets orally once daily; with a body weight of 76-90 kg were administered four 400 mg tablets orally once
- RHZE-RMZE: Participants were administered RHZE Day 1 to Day 2 and RMZE from Day 3 to Day 14.
  Rifampicin: Participants with body weight </= 50kg were administered one 450 mg tablet orally once daily; with body weight >50kg were administered one 600 mg tablet orally once daily.
  Isoniazid: Participants were administered three 100 mg tablets or one 300 mg tablet once daily.
  Pyrazinamide: Participants with a body weight of 40-55 kg were administered two 500 mg tablets orally once daily; with a body weight of 56-75 kg were administered three 500 mg tablets orally once daily; with a body weight of 76-90 kg were administered four 500 mg tablets orally once daily.
  Ethambutol: Participants with a body weight of 40-55 kg were administered two 400 mg tablets orally once daily; with a body weight of 56-75 kg were administered three 400 mg tablets orally once daily; with a body weight of 76-90 kg were administered four 400 mg tablets orally once daily.
  Moxifloxacin: one 400 mg tablet orally once a day.
- RZE-RZE: Participants were administered only RZE from Day 1 through Day 14. Rifampicin: Participants with body weight </= 50kg were administered one 450 mg tablet orally once daily; with body weight >50kg were administered one 600 mg tablet orally once daily.
  Pyrazinamide: Participants with a body weight of 40-55 kg were administered two 500 mg tablets orally once daily; with a body weight of 56-75 kg were administered three 500 mg tablets orally once daily; with a body weight of 76-90 kg were administered four 500 mg tablets orally once daily.
  Ethambutol: Participants with a body weight of 40-55 kg were administered two 400 mg tablets orally once daily; with a body weight of 56-75 kg were administered three 400 mg tablets orally once daily; with a body weight of 76-90 kg were administered four 400 mg tablets orally once daily.
Period: Overall Study
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Started | 18 | 17 | 16 | 18
Completed | 17 (1 participant who completed study but had insufficient sputum volume was excluded from the analyses) | 16 (1 participant who completed study but had insufficient sputum volume was excluded from the analyses) | 15 | 17
Not Completed | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Pre-entry overnight sputum< 10ML | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat: All enrolled 69 participants were included in the baseline characteristics.
Groups:
- RHZE-RHZE: Participants were administered RHZE from Day 1 to Day 14.
- RHZE-RZE: Participants were administered RHZE from Day 1 to Day 2, then RZE from Day 3 to Day 14.
- RHZE-RMZE: Participants were administered RHZE Day 1 to Day 2 and RMZE from Day 3 to Day 14.
- Total: Total of all reporting groups
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE | Total
Number analyzed (Participants) | 18 | 17 | 16 | 18 | 69
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28.5 [22 to 33] | 31 [30 to 35] | 33.5 [25.5 to 43] | 32 [21 to 44] | 31 [24 to 40]
Age, Customized [Count of Participants; unit: Participants]
  <20 | 2 | 0 | 1 | 1 | 4
  20-29 | 7 | 4 | 6 | 5 | 22
  30-39 | 5 | 11 | 2 | 5 | 23
  40-49 | 2 | 1 | 4 | 6 | 13
  50-59 | 2 | 1 | 3 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 3 | 12
  Male | 13 | 16 | 13 | 15 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 18 | 15 | 16 | 18 | 67
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 18 | 17 | 16 | 18 | 69
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Karnofsky score [Median (Full Range); unit: scores on a scale] — The karnofsky score was determined according to karnofsky performance scale. The scale ranged from 0 to 100, by 10. A higher value represents a better outcome.
  scores on a scale | 90 [80 to 100] | 90 [80 to 90] | 90 [80 to 90] | 90 [80 to 90] | 90 [80 to 100]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 18.5 [17.5 to 20.9] | 19.4 [17.5 to 20.4] | 19.8 [17.7 to 22.7] | 18.7 [16.8 to 20.4] | 18.9 [17.5 to 20.8]
HIV status [Number; unit: participants]
  HIV negative | 16 | 16 | 15 | 18 | 65
  HIV positive | 2 | 1 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Daily Decrease in log10 Transformed Colony-forming Unit (CFU) Counts Per ml Sputum From Baseline (Study Treatment Initiation) to Day 14
Description: The daily decrease was calculated as follows:
  EBA0-14(CFU)= [baseline log10 CFU/mL sputum (mean of log10 CFU/mL at pre-entry and day 0) - log10 CFU/mL at day 14]/14. For a CFU/ml count of 0, the log10 CFU/mL was set to 0.
  No formal statistical testing was conducted to compare the arms. Please refer to the explanation in the Protocol Section.
Time Frame: Pre-entry, Day 0 and Day 14
Population: Participants with qualified sputum samples who had results available at all time points specified in the time-frame
Measure: Median (Inter-Quartile Range); unit: log10 CFU/ mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 12 | 11 | 10 | 15
log10 CFU/ mL | 0.134 [0.078 to 0.167] | 0.096 [0.028 to 0.211] | 0.136 [0.090 to 0.169] | 0.119 [0.050 to 0.173]

2. Secondary Outcome: Daily Change in Time to Positivity (TTP) From Baseline (Study Treatment Initiation) to Day 14
Description: The daily change in TTP was calculated as follows:
  EBA0-14(TTP) = [baseline TTP (mean of TTP at pre-entry and day 0) - TTP at day 14]/14.
Time Frame: Pre-entry, Day 0 and Day 14
Population: Participants with qualified sputum samples who had results available at all time points specified in the time-frame
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 16
hours | -12 [-17 to -9] | -12 [-16 to -8] | -13 [-17 to -10] | -11 [-14 to -9]

3. Secondary Outcome: Daily Change in log10 Transformed Colony-forming Unit (CFU) Counts Per mL Sputum From Baseline (Study Treatment Initiation) to Day 2
Description: The daily change in log10 CFU/mL sputum was calculated as follows:
  EBA0-2(CFU) = (baseline log10 CFU/mL sputum (mean of log10 CFU/mL at pre-entry and day 0) - log10 CFU/mL at day 2)/2.
  For a CFU/mL count of 0, the log10 CFU/mL was set to 0.
Time Frame: Pre-entry, Day 0 and Day 2
Population: Participants with qualified sputum samples who had results available at all time points specified in the time-frame
Measure: Median (Inter-Quartile Range); unit: log10 CFU/ mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 12 | 13 | 12 | 12
log10 CFU/ mL | 0.255 [-0.037 to 0.519] | 0.385 [-0.050 to 0.475] | 0.111 [0.001 to 0.409] | 0.034 [-0.366 to 0.443]

4. Secondary Outcome: Daily Change in log10 Colony-forming Unit (CFU) Counts Per mL Sputum From Day 2 to Day 14
Description: The daily change in log10 CFU/mL sputum was calculated as follows:
  EBA2-14(CFU) = (log10 CFU/mL at day 2 - log10 CFU/mL at day 14)/12.
  For a CFU/mL count of 0, the log10 CFU/mL was set to 0.
Time Frame: Day 2 and day 14
Population: Participants with qualified sputum samples who had results available at all time points specified in the time-frame
Measure: Median (Inter-Quartile Range); unit: log10 CFU/ mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 10 | 11 | 11 | 11
log10 CFU/ mL | 0.143 [0.104 to 0.203] | 0.093 [0.010 to 0.171] | 0.123 [0.113 to 0.173] | 0.104 [0.065 to 0.277]

5. Secondary Outcome: Daily Change in Time to Positivity (TTP) From Baseline (Study Treatment Initiation) to Day 2
Description: The daily change in TTP was calculated as follows:
  EBA0-2(TTP) = (baseline TTP (mean of TTP at pre-entry and day 0) - TTP at day 2)/2.
Time Frame: Pre-entry, Day 0 and Day 2
Population: Participants with qualified sputum samples who had results available at all time points specified in the time-frame
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 16
hours | -31 [-44 to -22] | -30 [-44 to -15] | -29 [-35 to -18] | -25 [-28 to -18]

6. Secondary Outcome: Daily Change in Time to Positivity (TTP) From Day 2 to Day 14
Description: The daily change in TTP was calculated as follows:
  EBA2-14(TTP) = (TTP at day 2 - TTP at day 14)/12.
Time Frame: Day 2 and Day 14
Population: Participants with qualified sputum samples who had results available at all time points specified in the time-frame
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- RHZE-RMZE: Participants will be administered RHZE Day 1 to Day 2 and RMZE from Day 3 to Day 14.
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
hours | -9 [-12 to -6] | -9 [-13 to -6] | -12 [-14 to -8] | -9 [-12 to -7]

7. Secondary Outcome: Log10 Transformed Colony-forming Unit (CFU) Count Per mL From Sputum Samples at Baseline and Day 14
Description: The log10 CFU count per mL from sputum samples processed by standard method or decontaminated method.
Time Frame: Pre-entry, Day 0 and Day 14
Population: Participants with qualified sputum samples who had results available at least one time point specified in the time-frame
Measure: Median (Inter-Quartile Range); unit: log10 CFU/ mL
Groups:
- Standard Processing Method: The standard sputum processing method
- Decontaminated Processing Method: The decontaminated sputum processing method
Arm/Group | Standard Processing Method | Decontaminated Processing Method
Number analyzed (Participants) | 63 | 63
log10 CFU/ mL
  Pre-entry: number analyzed (Participants) | 54 | 54
  Pre-entry | 5.80 [5.16 to 6.76] | 5.89 [5.10 to 6.62]
  Day 0: number analyzed (Participants) | 51 | 56
  Day 0 | 5.68 [5.16 to 6.65] | 5.58 [5.02 to 6.41]
  Day 14: number analyzed (Participants) | 49 | 48
  Day 14 | 4.01 [3.34 to 4.60] | 3.74 [3.11 to 4.40]

8. Secondary Outcome: Correlation Between Time to Positivity (TTP) and log10 Transformed Colony-forming Unit (CFU) Counts Per mL
Description: Pearson correlation coefficient was used to examine the correlation between TTP and log10 CFU among all qualified samples obtained on study
Time Frame: Pre-entry, Day 0, Day 1, Day 2, Day 3, Day 5, Day 7, Day 9, Day 11 and Day 14
Population: as for outcome 7
Measure: Number; unit: correlation coefficient
Groups:
- Overall: Qualified samples from overall participants
Arm/Group | Overall
Number analyzed (Participants) | 63
correlation coefficient | -0.75

9. Secondary Outcome: Pharmacokinetic Parameter (PK) Area Under the Concentration-time Curve (AUC0-24hour) for Rifampicin (RIF)
Description: Pharmacokinetic Parameter Area Under the Concentration-time Curve (AUCs) of Rifampicin from 0 to 24 hours obtained at Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Rifampicin dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis
Measure: Median (Inter-Quartile Range); unit: h*ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
h*ng/mL
  RIF AUC0-24hour at Day 1 | 37358.8 [23946.7 to 70314.2] | 42062.6 [23048.7 to 77672.3] | 51434.1 [42018.3 to 69759.7] | 39294.0 [21282.6 to 55823.8]
  RIF AUC0-24hour at Day 14 | 31361.4 [15709.9 to 42480.9] | 27161.7 [14436.6 to 31522.2] | 26751.2 [16603.9 to 32635.8] | 30521.0 [20749.5 to 35307.8]

10. Secondary Outcome: Rifampicin PK Parameter Clearance (CL/F)
Description: Rifampicin PK parameter Clearance (CL/F) obtained Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Rifampicin dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis
Measure: Median (Inter-Quartile Range); unit: L/hour
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
L/hour
  RIF CL/F Day 1 | 14.0 [8.3 to 20.1] | 12.5 [7.7 to 26.0] | 10.5 [7.2 to 14.3] | 14.3 [9.2 to 21.1]
  RIF CL/F Day 14 | 18.0 [14.1 to 34.0] | 22.1 [14.3 to 31.2] | 21.5 [15.7 to 36.1] | 17.0 [14.7 to 22.0]

11. Secondary Outcome: Rifampicin PK Parameter Maximum Plasma Concentration (Cmax)
Description: Rifampicin PK parameter Parameter Maximum Plasma Concentration (Cmax) obtained Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Rifampicin dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
ng/mL
  RIF Cmax at Day 1 | 5565 [3600 to 7685] | 6060 [3200 to 9550] | 8660 [4520 to 10800] | 4880 [3370 to 7740]
  RIF Cmax at Day 14 | 7145 [3525 to 9055] | 6960 [3930 to 9020] | 7370 [4700 to 9580] | 8350 [5390 to 8970]

12. Secondary Outcome: Rifampicin PK Parameter Last Concentration (CLast)
Description: Rifampicin (RIF) PK parameter Last Concentration (CLast) obtained Day 1 and Day 14. The lower limit of quantification of the assay (LLOQ) for RIF was 40 ng/mL. The results below the lower limit of quantification were assigned as one-half the value of the LLOQ, which was 20 ng/mL.
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Rifampicin dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
ng/mL
  RIF CLast at Day 1 | 74.5 [20.0 to 232.0] | 20 [20 to 229] | 133 [20 to 288] | 20 [20 to 272]
  RIF CLast at Day 14 | 20 [20 to 20] | 20 [20 to 20] | 20 [20 to 20] | 20 [20 to 20]

13. Secondary Outcome: AUC0-24hour for Isoniazid (INH) at Day 1
Description: PK AUCs of Isoniazid (INH) from 0 to 24 hours obtained at Day 1
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Isoniazid dosing at Day 1
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis. The participants in the RZE-RZE arm did not receive INH from Day 1 through Day 14.
Measure: Median (Inter-Quartile Range); unit: h*ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE
Number analyzed (Participants) | 16 | 15 | 15
h*ng/mL | 10725.8 [6412.9 to 16492.5] | 7970.6 [4594.4 to 16101.7] | 7165.1 [4974.5 to 19045.0]

14. Secondary Outcome: Isoniazid PK Parameter CL/F at Day 1
Description: Isoniazid PK parameter CL/F obtained Day 1
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Isoniazid dosing at Day 1
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: L/hour
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE
Number analyzed (Participants) | 16 | 15 | 15
L/hour | 28.0 [18.3 to 49.6] | 37.6 [18.6 to 65.3] | 41.9 [21.0 to 60.6]

15. Secondary Outcome: Isoniazid PK Parameter Cmax at Day 1
Description: Isoniazid PK parameter Cmax obtained Day 1
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Isoniazid dosing at Day 1
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE
Number analyzed (Participants) | 16 | 15 | 15
ng/mL | 3165 [2315 to 4060] | 2920 [1530 to 3610] | 2760 [1760 to 4030]

16. Secondary Outcome: Isoniazid PK Parameter CLast at Day 1
Description: Isoniazid (INH) PK parameter CLast obtained Day 1. The lower limit of quantification of the assay (LLOQ) for INH was 100 ng/mL. The results below the lower limit of quantification were assigned as one-half the value of the LLOQ, which was 50 ng/mL.
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Isoniazid dosing at Day 1
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE
Number analyzed (Participants) | 16 | 15 | 15
ng/mL | 50 [50 to 50] | 50 [50 to 50] | 50 [50 to 50]

17. Secondary Outcome: AUC0-24hour for Isoniazid at Day 14
Description: PK AUCs of Isoniazid from 0 to 24 hours obtained at Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Isoniazid dosing at Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis. The participants in the RHZE-RZE and RHZE-RMZE arms did not receive INH from Day 3 through Day 14 and the participants in the RZE-RZE arm did not receive INH from Day 1 through Day 14.
Measure: Median (Inter-Quartile Range); unit: h*ng/mL
Arm/Group | RHZE-RHZE
Number analyzed (Participants) | 16
h*ng/mL | 9797.2 [6931.1 to 16355.9]

18. Secondary Outcome: Isoniazid PK Parameter CL/F at Day 14
Description: Isoniazid PK parameter CL/F obtained Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Isoniazid dosing at Day 14
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: L/hour
Arm/Group | RHZE-RHZE
Number analyzed (Participants) | 16
L/hour | 30.6 [18.4 to 46.0]

19. Secondary Outcome: Isoniazid PK Parameter Cmax at Day 14
Description: Isoniazid PK parameter Cmax obtained Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Isoniazid dosing at Day 14
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE
Number analyzed (Participants) | 16
ng/mL | 3130 [2485 to 3920]

20. Secondary Outcome: Isoniazid PK Parameter CLast at Day 14
Description: Isoniazid (INH) PK parameter CLast obtained Day 14. The lower limit of quantification of the assay (LLOQ) for INH was 100 ng/mL. The results below the lower limit of quantification were assigned as one-half the value of the LLOQ, which was 50 ng/mL.
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Isoniazid dosing at Day 14
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE
Number analyzed (Participants) | 16
ng/mL | 50 [50 to 50]

21. Secondary Outcome: AUC0-24hour for Pyrazinamide (PZA)
Description: PK AUCs of Pyrazinamide (PZA) from 0 to 24 hours obtained at Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Pyrazinamide dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Measure: Median (Inter-Quartile Range); unit: h*ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
h*ng/mL
  PZA AUC0-24hour at Day 1 | 301214.5 [243041.4 to 344110.0] | 255283.0 [204379.9 to 349309.1] | 292078.2 [249250.9 to 304794.0] | 272853.9 [217158.6 to 314465.1]
  PZA AUC0-24hour at Day 14 | 249879.1 [202652.1 to 319071.7] | 201389.7 [174896.2 to 280573.1] | 280071.0 [221878.7 to 312248.4] | 252276.8 [192061.9 to 307469.4]

22. Secondary Outcome: Pyrazinamide PK Parameter CL/F
Description: Pyrazinamide PK parameter CL/F obtained Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Pyrazinamide dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Measure: Median (Inter-Quartile Range); unit: L/hour
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
L/hour
  PZA CL/F Day 1 | 4.1 [3.3 to 5.0] | 4.8 [3.9 to 5.8] | 4.7 [3.4 to 5.2] | 4.2 [3.7 to 4.9]
  PZA CL/F Day 14 | 4.5 [4.0 to 6.5] | 5.4 [4.8 to 6.9] | 4.7 [3.9 to 5.3] | 4.7 [3.8 to 5.8]

23. Secondary Outcome: Pyrazinamide PK Parameter Cmax
Description: Pyrazinamide PK parameter Cmax obtained Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Pyrazinamide dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
ng/mL
  PZA Cmax at Day 1 | 27650 [24400 to 36550] | 27000 [20800 to 29100] | 28800 [23900 to 32600] | 25800 [24100 to 29000]
  PZA Cmax at Day 14 | 29300 [24950 to 34350] | 27000 [22900 to 31000] | 29300 [25500 to 33900] | 28000 [26300 to 31900]

24. Secondary Outcome: Pyrazinamide PK Parameter CLast
Description: Pyrazinamide PK parameter CLast obtained Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Pyrazinamide dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
ng/mL
  PZA CLast at Day 1 | 3370 [2320 to 5470] | 2850 [1500 to 5050] | 3130 [2570 to 3460] | 2710 [1930 to 3830]
  PZA CLast at Day 14 | 1955.0 [997.5 to 2735.0] | 1280 [909 to 3050] | 1790 [1450 to 2900] | 1770 [1270 to 2150]

25. Secondary Outcome: AUC0-24hour for Ethambutol (EMB)
Description: PK AUCs of Ethambutol (EMB) from 0 to 24 hours obtained at Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Ethambutol dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Measure: Median (Inter-Quartile Range); unit: h*ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
h*ng/mL
  EMB AUC0-24hour at Day 1 | 11918.8 [9783.4 to 12803.2] | 11145.8 [9336.6 to 14125.3] | 11322.4 [9549.6 to 13937.0] | 10716.8 [9381.2 to 13678.0]
  EMB AUC0-24hour at Day 14 | 16414.9 [13813.1 to 19637.1] | 16675.9 [12589.8 to 18585.1] | 15181.2 [14074.7 to 17338.1] | 16574.6 [13314.9 to 17422.2]

26. Secondary Outcome: Ethambutol PK Parameter CL/F
Description: Ethambutol PK parameter CL/F obtained Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Ethambutol dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Measure: Median (Inter-Quartile Range); unit: L/hour
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
L/hour
  EMB CL/F Day 1 | 93.6 [68.7 to 105.0] | 85.4 [73.9 to 97.1] | 83.8 [65.4 to 106.0] | 76.5 [73.9 to 89.8]
  EMB CL/F Day 14 | 57.9 [51.0 to 65.9] | 63.5 [53.5 to 72.0] | 56.8 [47.1 to 75.2] | 60.1 [52.4 to 64.4]

27. Secondary Outcome: Ethambutol PK Parameter Cmax
Description: Ethambutol PK parameter Cmax obtained Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Ethambutol dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
ng/mL
  EMB Cmax at Day 1 | 2650 [1745 to 2960] | 2040 [1840 to 2460] | 2470 [1790 to 3460] | 2220 [1900 to 2680]
  EMB Cmax at Day 14 | 2980 [2220 to 3525] | 3090 [2270 to 3370] | 2780 [2580 to 3220] | 2920 [2530 to 3250]

28. Secondary Outcome: Ethambutol PK Parameter CLast
Description: Ethambutol PK parameter CLast obtained Day 1 and Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Ethambutol dosing at Day 1 and Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
Number analyzed (Participants) | 16 | 15 | 15 | 17
ng/mL
  EMB CLast at Day 1 | 86.5 [40.0 to 106.5] | 85 [40 to 107] | 40 [40 to 94] | 86 [40 to 95]
  EMB CLast at Day 14 | 205.0 [167.0 to 235.5] | 176 [159 to 208] | 164 [136 to 199] | 159 [134 to 204]

29. Secondary Outcome: AUC0-24hour for Moxifloxacin (Mox) at Day 14
Description: PK AUCs of Moxiflozacin (Mox) from 0 to 24 hours obtained at Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Moxifloxacin dosing at Day 14
Population: 63 with qualified samples were included in the primary and secondary analyses including PK analysis. Only the participants in the RHZE-RMZE arm received Mox from Day 3 through Day 14
Measure: Median (Inter-Quartile Range); unit: h*ng/mL
Arm/Group | RHZE-RMZE
Number analyzed (Participants) | 15
h*ng/mL | 22498.4 [21012.8 to 23318.5]

30. Secondary Outcome: Moxifloxacin PK Parameter CL/F at Day 14
Description: Moxifloxacin PK parameter CL/F obtained Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Moxifloxacin dosing at Day 14
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: L/hour
Arm/Group | RHZE-RMZE
Number analyzed (Participants) | 15
L/hour | 17.8 [17.2 to 19.0]

31. Secondary Outcome: Moxifloxacin PK Parameter Cmax at Day 14
Description: Moxifloxacin PK parameter Cmax obtained Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Moxifloxacin dosing at Day 14
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RMZE
Number analyzed (Participants) | 15
ng/mL | 3010 [2710 to 3500]

32. Secondary Outcome: Moxifloxacin PK Parameter CLast at Day 14
Description: Moxifloxacin PK parameter CLast obtained Day 14
Time Frame: -0.5 hour (pre-dose), 1, 2, 3, 5, 7, 10, 12 and 24 hours after Moxifloxacin dosing at Day 14
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | RHZE-RMZE
Number analyzed (Participants) | 15
ng/mL | 178 [150 to 217]

ADVERSE EVENTS:
Time Frame: From treatment dispensation to study discontinuation. The duration of the study was 29 days.
Description: The protocol required reporting of all new diagnoses and new signs and symptoms and laboratory abnormalities of >=Grade 2. The DAIDS Adverse Event (AE) Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used for grading of AEs. Expedited adverse event reporting followed Version 2.0 of the DAIDS Expedited Adverse Event Manual.
Arm/Group | RHZE-RHZE | RHZE-RZE | RHZE-RMZE | RZE-RZE
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/17 | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/17 | 1/16 | 0/18
Other Adverse Events (participants affected / at risk) | 6/18 | 5/17 | 3/16 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RHZE-RHZE (N=18) | RHZE-RZE (N=17) | RHZE-RMZE (N=16) | RZE-RZE (N=18)
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RHZE-RHZE (N=18) | RHZE-RZE (N=17) | RHZE-RMZE (N=16) | RZE-RZE (N=18)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.